CLINICAL TRIAL: NCT06209827
Title: Effectiveness of a Multidisciplinary Intervention in the Reduction of Benzodiazepine Prescriptions: A Cluster Controlled Trial
Brief Title: Effectiveness of a Community Intervention in the Chronic Use of Benzodiazepines: (BENZOSTOPJUNTOS)
Acronym: BENZOSTOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andalusian Health Service (Other Government)
Collaborators: Andalusian School of Public Health (Other Government)
Responsible Party: Principal Investigator, Ingrid Ferrer López, Principal Investigator. Primary Care Pharmacist. Pharm.G, Ph.D. Clinical management unit Primary care pharmacy Seville.Andalusian Health Service, Andalusian Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IFLBZD16
Record Dates: First submitted 2024-01-06; First posted 2024-01-18 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Inappropriate Prescribing
Keywords: Benzodiazepine; Medication overuse.; Inappropriate Prescribing
MeSH Terms: conditions — Prescription Drug Overuse | interventions — Methods

STUDY DESIGN:
Intervention Model Description: cluster-randomized, parallel-group trial in which health centres were the units of randomization and patients were the units of analysis
Who Masked: Outcomes Assessor
Masking Description: Data collector was not involved in outcomes assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention for reducing benzodiazepines long-term use. (Experimental): It included the multiple components as follows:
  (i) an exchange discussion with the patient describing the advantages, disadvantages and alternatives of benzodiazepines use and a tapering protocol with the support of educational material, (ii) the offer of a brief, if necessary, consultation with the family doctor, and (iii) a letter addressed to the patient supported by scientific societies.
  Interventions: Behavioral: Intervention for reducing benzodiazepines long-term use.
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Intervention for reducing benzodiazepines long-term use. — Comprehensive, multicomponent intervention utilizing education and support for benzodiazepines.
  Family doctor, nurse, community pharmacist and social workers: carried out informative discussion with the patient with by providing educational material. They informed patients about the advantages, disadvantages and alternatives to benzodiazepines including a descending benzodiazepines schedule to minimize withdrawal symptoms. It briefly explained the professionals' concerns about the continued use of benzodiazepines and offers possible solutions.
  If the patient requested a withdrawal, he/she was referred to the doctor.
  Arms: Intervention for reducing benzodiazepines long-term use.

SUMMARY:
This study aimed to assess the effectiveness of a comprehensive, multicomponent intervention utilizing education and support for Benzodiazepines withdrawal compared to standard care.

DETAILED DESCRIPTION:
The excessive use of benzodiazepines (BZDs) presents significant health concerns and high healthcare costs, particularly in Spain, where usage rates are among the highest globally. In Andalusian, over a 10% of the population use BZDs long-term, prompting the need for safe and effective reduction strategies.

This study aimed to assess the effectiveness of a comprehensive, multicomponent intervention utilizing education and support for BZD withdrawal compared to standard care.

The intervention involved educational discussions, consultations with health professionals, and letters supported by multiple scientific societies.

ELIGIBILITY:
Inclusion Criteria:

* users of health centre's with more than 4 weeks of benzodiazepines use.
* users of health centre's over 18 years of age.

Exclusion Criteria:

* users of health centre's with mental disorder.
* users of health centre's terminal.
* users of health centre's with alcohol dependence.
* users of health centre's with dementia.
* users of health centre's who had intellectual disabilities.
* users of health centre's unable to cooperate with the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of dispensing of benzodiazepines. | 3.5 years
  Number of dispensing of benzodiazepines, measured at the level of the participant.

SECONDARY OUTCOMES:
Knowledge | 6 months
  Knowledge: Empower questionary, measured at the level of the participant.
Life Quality | 6 months
  Quality of life:Functional Status Measurement Sheets by coop World Organisation of Family Doctors (COOP/ WONCA):
  The six COOP-WONCA Charts are described by vignettes and measured at the level of the participant: physical fitness, feelings, daily activities, social activities, change in health and overall health.
  WONCA: World Organisation of Family Doctors

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Ferrer López, Ph.D, Principal Investigator — SAS
Locations (1):
- Ingrid Ferrer López, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferrer Lopez I, Olry de Labry-Lima A, Gutierrez-Valencia A, Garcia Bermudez E, Atienza Martin F, Morente AG, Murillo Fernandez MD, Sanchez Canete Y, Bermudez-Tamayo C. Risk perception, attitudes, and quality of life in a multicomponent benzodiazepine deprescription strategy. Explor Res Clin Soc Pharm. 2025 Sep 30;20:100666. doi: 10.1016/j.rcsop.2025.100666. eCollection 2025 Dec. PMID 41142506